CLINICAL TRIAL: NCT02838914
Title: Assessment of Reconstruction and Inverse Reconstruction in Right Atrium by by Multimodal Echocardiographic Techniques for Atrial Fibrillation Patients Before and After Radiofrequency Ablation
Brief Title: Assessment of Reconstruction and Inverse Reconstruction in Right Atrium by Multimodal Echocardiographic Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yi Yu, vice professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-16-006
Record Dates: First submitted 2016-04-15; First posted 2016-07-20 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Right atrium; Echocardiography; Remodeling
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients with AF (Experimental): Before radiofrequency ablation (RFCA)
  Interventions: Procedure: radiofrequency ablation (RFCA)
- Assigned Comparisons (Experimental): After radiofrequency ablation (RFCA)
  Interventions: Procedure: radiofrequency ablation (RFCA)

INTERVENTIONS:
Procedure: radiofrequency ablation (RFCA) — Patients undergo radiofrequency ablation (RFCA)

SUMMARY:
The purpose of the study is to assess the reconstruction and inverse reconstruction in right atrium by speckle tracking echocardiography combined with real-time three dimensional echocardiography for atrial fibrillation patients before and after radiofrequency ablation (RFCA)

DETAILED DESCRIPTION:
The prevalence of atrial fibrillation (AF) has increased in recent years. The construction and function of right atrium haven't shown clearly before and after radiofrequency ablation (RFCA).The purpose of the study is to investigate whether RFCA can lead to inverse reconstruction of right atrium for atrial fibrillation patients, which diagnosing by speckle tracking echocardiography combined with real-time three dimensional echocardiography. All patients will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. With a history of paroxysmal Af (PAF) and PAF record within 6 months prior to ablation, confirming at least one of the following findings: AF lasting for ≥30 s recorded in Holter or 12-lead ECG.
2. No response to more than one antiarrhythmic drug, or unwilling to receive longterm drug treatment.
3. Can provide informed consent form expressing willingness to participate in the study and comply with follow-up tests and evaluation procedures.
4. Aged 18-80 years.

Exclusion Criteria:

1. With acute diseases, such as acute phase after myocardial infarction (within 3 months), within 3 months after acute heart failure or new cerebral infarction;
2. In the list of heart transplantation;
3. Expected survival less than 1 year;
4. With other hemorrhagic diseases and anticoagulant therapy is not allowed;
5. Thrombosis in left atrium;
6. Heart failure, New York Heart Association(NYHA) III/IV or eject fraction(EF)<40%;
7. Patients with uncontrolled cancer;
8. Significant hepatic or renal impairment (and/or alanine transaminase(ALT) or Aspartate transaminase(AST) >2 times upper limit of normal, creatinine clearance rate(CCr)<50%);
9. Previous catheter radiofrequency ablation for AF or cardiac surgery;
10. Pregnant and lactating women, women who plan to become pregnant, or women of child bearing age not using reliable contraceptive measures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Remodeling in right atrium measured by speckle tracking echocardiography combined with real-time three dimensional echocardiography in AF patients | In one week before RFCA

SECONDARY OUTCOMES:
Remodeling in right atrium measured by speckle tracking echocardiography combined with real-time three dimensional echocardiography in AF patients | In one week after RFCA
Inverse reconstruction in right atrium measured by speckle tracking echocardiography combined with real-time three dimensional echocardiography in AF patients | At three months after RFCA
Inverse reconstruction in right atrium measured by speckle tracking echocardiography combined with real-time three dimensional echocardiography in AF patients | At six months after RFCA
Adverse event that is related to RFCA, such as the incidence of cardiac tamponade (%) was obtained by echocardiography | In one week after RFCA

OTHER OUTCOMES:
Adverse events that are related to RFCA, such as the incidence of pulmonary vein stenosis(%) and embolism(%) were obtained by CT | At six months after RFCA

CONTACTS AND LOCATIONS:
Overall Officials: Kun Sun, M.D.;Ph.D., Principal Investigator — Department of Ultrasound, Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Xinhua Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thihalolipavan S, Morin DP. Atrial fibrillation and congestive heart failure. Heart Fail Clin. 2014 Apr;10(2):305-18. doi: 10.1016/j.hfc.2013.12.005. Epub 2014 Feb 4. PMID 24656107
- [Result] Extramiana F, Maison-Blanche P. Stroke and atrial fibrillation: where to go from here? Stroke. 2015 Mar;46(3):605-7. doi: 10.1161/STROKEAHA.114.007809. Epub 2015 Jan 29. No abstract available. PMID 25634002
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Result] Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH; ESC Committee for Practice Guidelines. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Europace. 2010 Oct;12(10):1360-420. doi: 10.1093/europace/euq350. No abstract available. PMID 20876603
- [Result] Rondano E, Dell'Era G, De Luca G, Piccinino C, Bellomo G, Marino PN. Left atrial asynchrony is a major predictor of 1-year recurrence of atrial fibrillation after electrical cardioversion. J Cardiovasc Med (Hagerstown). 2010 Jul;11(7):499-506. doi: 10.2459/JCM.0b013e32833757b5. PMID 20445461
- [Result] Wang Z, Tan H, Zhong M, Jiang G, Zhang Y, Zhang W. Strain rate imaging for noninvasive functional quantification of the left atrium in hypertensive patients with paroxysmal atrial fibrillation. Cardiology. 2008;109(1):15-24. doi: 10.1159/000105322. Epub 2007 Jul 10. PMID 17627105
- [Result] Lee YS, Hyun DW, Jung BC, Cho YK, Lee SH, Shin DG, Park HS, Han SW, Kim YN; KTK Cardiac Electrophysiology Working Group. Left atrial volume index as a predictor for occurrence of atrial fibrillation after ablation of typical atrial flutter. J Cardiol. 2010 Nov;56(3):348-53. doi: 10.1016/j.jjcc.2010.07.006. PMID 20889311
- [Result] Muller H, Reverdin S, Burri H, Shah D, Lerch R. Measurement of left and right atrial volume in patients undergoing ablation for atrial arrhythmias: comparison of a manual versus semiautomatic algorithm of real time 3D echocardiography. Echocardiography. 2014 Apr;31(4):499-507. doi: 10.1111/echo.12391. Epub 2013 Oct 15. PMID 24128369
- [Result] Peluso D, Badano LP, Muraru D, Dal Bianco L, Cucchini U, Kocabay G, Kovacs A, Casablanca S, Iliceto S. Right atrial size and function assessed with three-dimensional and speckle-tracking echocardiography in 200 healthy volunteers. Eur Heart J Cardiovasc Imaging. 2013 Nov;14(11):1106-14. doi: 10.1093/ehjci/jet024. Epub 2013 Feb 19. PMID 23423966
- [Result] Marwick TH, Leano RL, Brown J, Sun JP, Hoffmann R, Lysyansky P, Becker M, Thomas JD. Myocardial strain measurement with 2-dimensional speckle-tracking echocardiography: definition of normal range. JACC Cardiovasc Imaging. 2009 Jan;2(1):80-4. doi: 10.1016/j.jcmg.2007.12.007. PMID 19356538
- [Result] Reant P, Labrousse L, Lafitte S, Bordachar P, Pillois X, Tariosse L, Bonoron-Adele S, Padois P, Deville C, Roudaut R, Dos Santos P. Experimental validation of circumferential, longitudinal, and radial 2-dimensional strain during dobutamine stress echocardiography in ischemic conditions. J Am Coll Cardiol. 2008 Jan 15;51(2):149-57. doi: 10.1016/j.jacc.2007.07.088. PMID 18191740
- [Result] Mor-Avi V, Lang RM, Badano LP, Belohlavek M, Cardim NM, Derumeaux G, Galderisi M, Marwick T, Nagueh SF, Sengupta PP, Sicari R, Smiseth OA, Smulevitz B, Takeuchi M, Thomas JD, Vannan M, Voigt JU, Zamorano JL. Current and evolving echocardiographic techniques for the quantitative evaluation of cardiac mechanics: ASE/EAE consensus statement on methodology and indications endorsed by the Japanese Society of Echocardiography. Eur J Echocardiogr. 2011 Mar;12(3):167-205. doi: 10.1093/ejechocard/jer021. PMID 21385887
- [Result] Mirza M, Caracciolo G, Khan U, Mori N, Saha SK, Srivathsan K, Altemose G, Scott L, Sengupta P, Jahangir A. Left atrial reservoir function predicts atrial fibrillation recurrence after catheter ablation: a two-dimensional speckle strain study. J Interv Card Electrophysiol. 2011 Sep;31(3):197-206. doi: 10.1007/s10840-011-9560-6. Epub 2011 Mar 22. PMID 21424845
- [Result] Puwanant S, Park M, Popovic ZB, Tang WH, Farha S, George D, Sharp J, Puntawangkoon J, Loyd JE, Erzurum SC, Thomas JD. Ventricular geometry, strain, and rotational mechanics in pulmonary hypertension. Circulation. 2010 Jan 19;121(2):259-66. doi: 10.1161/CIRCULATIONAHA.108.844340. Epub 2010 Jan 4. PMID 20048214